CLINICAL TRIAL: NCT03630250
Title: Challenge of the Nasopharynx With Neisseria Lactamica Expressing the Meningococcal Protein Neisseria Adhesin A (NadA)
Acronym: NadA-Lac4
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NadA-Lac4
Record Dates: First submitted 2018-08-03; First posted 2018-08-14 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Meningitis, Bacterial; Neisseria Infection
Keywords: meningitis; GMO
MeSH Terms: conditions — Meningitis, Bacterial; Meningitis

STUDY DESIGN:
Intervention Model Description: Cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Challenge Volunteer - 4BN1 (Experimental): Volunteers will be given a choice of which version of the GM N. lactamica they would like to be given (4BN1 or 4YB2).
  On Day 0 Challenge volunteers will be asked to lie on their back, 0.5 mL of fluid containing a carefully measured amount of 4BN1 will be dripped slowly into each nostril. The volunteer will be able to breathe through their mouth during the procedure. Volunteers will be asked to remain lying down for 15 minutes. This will be performed only once.
  Volunteers will then be admitted to the NIHR Southampton CRF for 5 days. Challenge volunteers will then be asked to return for follow up visits on Day 7, 10, 14, 28, 56 90 & 92.
  A single dose of an antibiotic (Ciprofloxacin) will be administered on day 90 regardless of colonisation with modified N. lactamica 4BN1.
  Interventions: Biological: N. lactamica
- Contact Volunteer (No Intervention): Contact volunteers are those volunteers whose partner/spouse is a Challenge volunteer. Investigators will monitor Contact volunteers to collect information about transmission. A single dose of an antibiotic (Ciprofloxacin) will be administered on Day 90 regardless of colonisation with modified N. lactamica.
- Challenge Volunteer - 4YB2 (Experimental): Volunteers will be given a choice of which version of the GM N. lactamica they would like to be given (4BN1 or 4YB2).
  On Day 0 Challenge volunteers will be asked to lie on their back, 0.5 mL of fluid containing a carefully measured amount of 4YB2 will be dripped slowly into each nostril. The volunteer will be able to breathe through their mouth during the procedure. Volunteers will be asked to remain lying down for 15 minutes. This will be performed only once.
  Volunteers will then be admitted to the NIHR Southampton CRF for 5 days. Challenge volunteers will then be asked to return for follow up visits on Day 7, 10, 14, 28, 56 90 & 92.
  A single dose of an antibiotic (Ciprofloxacin) will be administered on day 90 regardless of colonisation with modified N. lactamica 4YB2
  Interventions: Biological: N. lactamica

INTERVENTIONS:
Biological: N. lactamica — Genetically modified N. lactamica
  Arms: Challenge Volunteer - 4BN1; Challenge Volunteer - 4YB2

SUMMARY:
This study is part of a research programme that aims to improve ways of protecting people from serious illnesses such as meningitis and sepsis caused by a bacterium called Neisseria meningitidis (N. meningitidis), using a closely related but harmless bacterium called Neisseria lactamica (N. lactamica). Investigators have previously given nose drops containing N. lactamica to over 350 volunteers - this is known as inoculation. In these studies the investigators have shown that they can cause colonisation of many inoculated volunteers (35-60%) with N. lactamica. Colonisation is when bacteria survive on or in a person without causing any illness or disease. N. lactamica specifically colonises the nose and throat. Investigators have also shown that colonisation with N. lactamica results in an immune (antibody) response.

In this study investigators will be using a genetically modified version of N. lactamica which contains a single gene from N. meningitides. It is anticipated that the presence of this gene will change the number of people who are colonised and how long people remain colonised for, as well as causing them to produce an immune response to N. meningitides.

The purpose of this study are to prove that inoculation with this modified N. lactamica does not cause any symptoms or illness, and to analyse the immune response produced in healthy volunteers.

DETAILED DESCRIPTION:
The NadA protein is one of the 4 strongly immunogenic components of the 4CMenB vaccine against serogroup B meningococcal disease (Bexsero) and has been demonstrated to be immunogenic in terms of generating serum bactericidal antibodies against N. meningitides strains that express the cognate NadA. Furthermore, University students vaccinated with Bexsero exhibit moderately reduced acquisition of nasopharyngeal carriage of N. meningitidis over the course of 12 months after vaccination. These studies imply that NadA expression by N. meningitidis may induce systemic and mucosal immunity to NadA during carriage, and that immunity directed against NadA may protect against colonisation by N. meningitidis. A greater understanding of the mucosal immune mechanisms of protection against pathobionts is essential for design of more effective and long lasting vaccines in the future. Then direct way to do this would be experimental human challenge with N. meningitidis but this carries potential hazard. As N. lactamica human challenge has shown to be safe, an alternative technique to investigate mucosal immunity to meningococcal antigens such as NadA will utilise Genetically Modified Organisms (GMOs) such as the one described here. Two strains of genetically modified N. lactamica will be used in this study, both of which have been derived from a beta-D-galactosidase (lacZ)-deficient mutant strain of N. lactamica Y92-1009 (△lacZ). This mutant can be differentiated from wild type bacteria when grown on the chromogenic substrate, X-gal. Both Genetically modified (GM) strains have demonstrated to remain acutely susceptible to killing by normal human serum and retain sensitivity to the front-line antibiotics used clinically to treat meningococcal disease (rifampicin, ciprofloxacin and ceftriaxone). The efficacy of ciprofloxacin to clear N. lactamica carriage is likely to similar as for N. meningitidis, as the organism is extremely sensitive to this antibiotic. Ciprofloxacin has been effective in clearing N. lactamica carriage within 24 hours in 100% of 4 individuals experimentally colonised in an ongoing human challenge study with wild type N. lactamica (unpublished data).

ELIGIBILITY:
Inclusion Criteria:

The challenge volunteer must satisfy all the following inclusion criteria to be eligible for the study:

* Healthy adults aged 18 to 45 years inclusive on the day of enrolment
* Fully conversant in the English language
* Able and willing (in the investigator's opinion) to comply with all study requirements
* Provide written informed consent to participate in the trial
* Provide written agreement to abide by infection control guidelines including agreement to abstain from intimate contact with any individual other than one declared and consented bedroom contact during the study period
* Provide written consent to allow the study team to discuss the volunteer's medical history with the General Practitioner
* Written informed contact volunteer consent provided by any bedroom contact
* Agreement to be admitted to Southampton NIHR-CRF for 4.5 days following inoculation
* For females only, willingness to practice continuous effective contraception (see below) during the study and a negative pregnancy test on the day(s) of screening and inoculation
* Able to correctly answer all questions in the pre-consent and infection control questionnaires
* Agreement to take antibiotic eradication therapy according to the study protocol
* TOPS registration completed and no conflict found

Exclusion Criteria:

The challenge volunteer may not enter the study if any of the following criteria apply:

* Current active smokers defined as having smoked a cigarette or cigar in the last four weeks
* N. lactamica or N. meningitidis detected on throat swab or nasal wash taken at screening or at the pre-challenge visit
* Individuals who have a current infection at the time of inoculation
* Individuals who have been involved in other clinical trials involving receipt of an investigational product over the last 12 weeks or if there is planned use of an investigational product during the study period
* Individuals who have previously been involved in clinical trials investigating meningococcal vaccines or experimental challenge with N. lactamica
* Individuals who have received one or more doses of the meningococcus B vaccine Bexsero
* Use of systemic antibiotics within the period 30 days prior to the challenge
* Any confirmed or suspected immunosuppressive or immune-deficient state, including HIV infection; malignancy, asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (topical steroids are allowed)
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* History of allergic disease or reactions likely to be exacerbated by any component of the inoculum
* Contraindications to the use of ciprofloxacin, specifically a history of epilepsy, prolonged QT interval, hypersensitivity to quinolones or a history of tendon disorders related to quinolone use
* Contraindications to the use of ceftriaxone, specifically hypersensitivity to any cephalosporins
* Any clinically significant abnormal finding on clinical examination or screening investigations. In the event of abnormal test results, confirmatory repeat tests will be requested.
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data, for example recent surgery to the nasopharynx
* Occupational, household or intimate contact with immunosuppressed persons, specifically HIV infection with a CD4 count <200 cells/mm3; asplenia; any malignancy, recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (topical steroids are allowed)
* Occupational or household contact with children under 5 years or an older child with a tendency to co-sleep with the volunteer
* Pregnancy, lactation or intention to become pregnant during the study
* Inability of the study team to contact the volunteer's GP to confirm medical history and safety to participate

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Establish the effect of the nasal inoculation of healthy volunteers with a genetically modified strain of Neisseria lactamica expressing NadA by measuring respiratory rate. | Up to volunteer visit Day 4
  Volunteers are admitted to the NIHR Southampton CRF and closely observed by trained medical members for any potential effects. Respiratory rate (breaths per minute) will be measured and compared with baseline measurements. A consistent increase in respiratory rate could indicate ill health and potential disease. A study doctor will review each participant twice a day for the duration of the inpatient stay.
Establish the effect of the nasal inoculation of healthy volunteers with a genetically modified strain of Neisseria lactamica expressing NadA by measuring body temperature. | Up to volunteer visit Day 4
  Volunteers are admitted to the NIHR Southampton CRF and closely observed by trained medical members for any potential effects. Body temperature (degrees Celsius) will be measured and compared with baseline measurements. A constant increase in body temperature could indicate ill health and potential disease. A study doctor will review each participant twice a day for the duration of the inpatient stay.
Establish the effect of the nasal inoculation of healthy volunteers with a genetically modified strain of Neisseria lactamica expressing NadA by measuring heart rate. | Up to volunteer visit Day 4
  Volunteers are admitted to the NIHR Southampton CRF and closely observed by trained medical members for any potential effects. Heart rate (beats per minute) will be measured and compared with baseline measurements. An increase in heart rate could indicate ill health and potential disease. A study doctor will review each participant twice a day for the duration of the inpatient stay.
Establish the effect of the nasal inoculation of healthy volunteers with a genetically modified strain of Neisseria lactamica expressing NadA by measuring blood pressure. | Up to volunteer visit Day 4
  Volunteers are admitted to the NIHR Southampton CRF and closely observed by trained medical members for any potential effects. Blood pressure (mmHg) will be measured and compared with baseline measurements. An increase in blood pressure could indicate ill health and potential disease. A study doctor will review each participant twice a day for the duration of the inpatient stay.

SECONDARY OUTCOMES:
To measure the NadA specific immunity in healthy volunteers following nasal inoculation with Neisseria lactamica expressing NadA | Up to volunteer visit Day 92
  Colonisation by Neisseria lactamica has previously shown to elicit a mucosal antibody response. Saliva samples will be collected from volunteers and antibody levels (µg/mL) specific to NadA pre and post inoculation will be measured to confirm if there is an increase. Those volunteers successfully colonised are hypothesised to show an increase in antibody production.

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Read, Principal Investigator — University of Southampton
Locations (1):
- NIHR Southampton Clinical Research Facility, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Laver JR, Hughes SE, Read RC. Neisserial Molecular Adaptations to the Nasopharyngeal Niche. Adv Microb Physiol. 2015;66:323-55. doi: 10.1016/bs.ampbs.2015.05.001. Epub 2015 May 30. PMID 26210107
- [Background] Deasy AM, Guccione E, Dale AP, Andrews N, Evans CM, Bennett JS, Bratcher HB, Maiden MC, Gorringe AR, Read RC. Nasal Inoculation of the Commensal Neisseria lactamica Inhibits Carriage of Neisseria meningitidis by Young Adults: A Controlled Human Infection Study. Clin Infect Dis. 2015 May 15;60(10):1512-20. doi: 10.1093/cid/civ098. Epub 2015 Mar 25. PMID 25814628
- [Background] Evans CM, Pratt CB, Matheson M, Vaughan TE, Findlow J, Borrow R, Gorringe AR, Read RC. Nasopharyngeal colonization by Neisseria lactamica and induction of protective immunity against Neisseria meningitidis. Clin Infect Dis. 2011 Jan 1;52(1):70-7. doi: 10.1093/cid/ciq065. PMID 21148522
- [Derived] Gbesemete D, Laver JR, de Graaf H, Ibrahim M, Vaughan A, Faust S, Gorringe A, Read RC. Protocol for a controlled human infection with genetically modified Neisseria lactamica expressing the meningococcal vaccine antigen NadA: a potent new technique for experimental medicine. BMJ Open. 2019 May 1;9(4):e026544. doi: 10.1136/bmjopen-2018-026544. PMID 31048443